CLINICAL TRIAL: NCT04597944
Title: Evaluation of the Efficacy of Kallikrein Inhibition by Lanadelumab for Patients With Bradykinin Angioedema: a Cohort Study
Brief Title: Lanadelumab in Bradykinin Angioedema
Acronym: KALAN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.187; 2020-A01528-31 (Other: ID RCB)
Record Dates: First submitted 2020-09-14; First posted 2020-10-22 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Angioedema
Keywords: Kallikrein, Kininogen, Bradykinin, Lanadelumab
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Hereditary or Acquired Angioedema: Participants older than 18 years that are diagnosed with Hereditary or Acquired Angioedema and treated by lanadelumab.

SUMMARY:
A multicenter observational study aiming to evaluate the efficacy of kallikrein inhibition by lanadelumab in patients with bradykinin- angioedema

DETAILED DESCRIPTION:
The bradykinin-angioedema (AE-BK) is characterized by recurrent and unpredictable episodes of swelling; it can be disabling and disfiguring and the attacks affecting the larynx can be life-threatening.

The clinical symptoms depend on accumulation of bradykinin (BK), a vasoactive peptide responsible for vasodilation and increase of vascular leakage. BK formation depends on activation of the kallikrein-kinin cascade leading to uncontrolled generation of plasma kallikrein and subsequent proteolysis of high molecular-weight kininogen (HK).

Lanadelumab is a fully human monoclonal antibody inhibitor of plasma kallikrein, thereby preventing BK production; it represents an attractive therapeutic strategy for BK-AE prophylaxis.

The aim of this study is to evaluate the kallikrein inhibition by assessing the levels of cleaved HK and the immunogenicity of the lanadelumab.

ELIGIBILITY:
Inclusion Criteria:

* Male/female >18 years old
* Patient with hereditary or acquired angioedema
* Patient treated by lanadelumab
* Patient whose the biological explorations have been carried out or will be carried out at Laboratory of Immunology of CHUGA
* Informed consent is obtained from the participant

Exclusion Criteria:

* Absence of biological material at T0 and M3 (stored for routine analysis)
* Person under guardianship or curatorship
* Female who is pregnant, nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hereditary or Acquired Angiodema
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of the kallikrein inhibition by lanadelumab in patients with bradykinin-angioedema | 3 months
  Levels of cleaved HK measured by Western Blot

SECONDARY OUTCOMES:
Evaluation of the efficacy of kallikrein inhibition by lanadelumab in patients with bradykinin-angioedema between T0 and the others visits | Day 7; 6, 12 and if possible 24 months
  Levels of cleaved HK as measured by Western Blot Ratio Day 7/ Day 0, Ratio Month 6/ Day 0, Ratio Month 12/ Day (and if possible Month 24/ Day 0) of the levels of cleaved HK as measured by Western Blot
  - SE2: antidrug antibodies in the sera of patients at Months 3, 6, 12 (and if possible Month 24).
Immunogenicity of lanadelumab | Months 3, 6, 12 (and 24 if possible)
  Levels of antidrug antibodies in the sera of patients
Evaluation of therapeutic escape | Months 3, 6, 12 and if possible 24
  Increase/absence of decrease of the number of attacks during lanadelumab administration

CONTACTS AND LOCATIONS:
Overall Officials: Federica DEFENDI, Principal Investigator — Grenoble Alpes University Hospital
Locations (2):
- France (2):
  - Chu Grenoble Alpes, Grenoble
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No